CLINICAL TRIAL: NCT04940260
Title: Long Term Renal Outcome in Preeclampsia : Role of sFlt-1 / PlGF and Endoglin
Brief Title: Soluble Factors and Renal Outcome in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 082/61
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Preeclampsia; Renal Function
MeSH Terms: conditions — Pre-Eclampsia | interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Renal function — measure eGFR at one year post partum
Diagnostic Test: proteinuria — measure urine protein creatinine ratio at one year postpartum

SUMMARY:
Preeclampsia (PE) is an important complication of pregnancy and can lead to chronic kidney disease by causing endothelial damage and podocyte loss, Soluble forms-like tyrosine kinase-1 (sFlt-1), placental growth factor (PlGF), sFlt1 / PlGF ratio and endoglin are the biomarkers for the differential diagnosis of preeclampsia and other diseases. We aim to explore the correlation of these biomarkers with long term renal function, blood pressure and urine albumin creatinine ratio (UACR) in PE patients.

DETAILED DESCRIPTION:
This is prospective observational study.Study subjects are pregnant women aged more than 18 years more than 24 weeks of gestation who were diagnosed and classified as preeclampsia or gestational hypertension by the criteria recommends by the American College of Obstetricians and Gynecologists (ACOG).14

Severe preeclampsia will be diagnosed by:

* A systolic/diastolic blood pressure ≥ 140 mmHg occurring on two occasions at least 4 hours apart after 20 weeks of gestation a women whose blood pressure has previously been normal
* Proteinuria with excretion of 0.3 gm or more of protein in a 24 hour urine specimen or urine dipstick results of at least 1+(30 mg per deciliter) on two occasions The exclusion criteria were chronic hypertension before pregnancy ,chronic kidney disease according to KDIGO criteria15 ,twin pregnancies,underlying diabetes mellitus .Of the 42 women enrolled in this trial,we excluded 2 patients who had twin pregnancies and history of diabetes mellitus. Eight women were lost to follow up. The remaining 32 patients completed the study.

Data collection and Laboratory Measurements Baseline demographic and clinical data will be recorded as follows: age, gestational age, blood pressure, medication history, parity. Laboratory data included complete blood count, blood urea nitrogen (BUN), creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), albumin, alkaline phosphate, lactate dehydrogenase (LDH), 24 -hour urine protein excretion and random urine protein-creatinine ratio. Enzyme-linked immunosorbent assay (ELISAs) for human soluble endoglin, SFlt1, and free PIGF will be conducted in duplicate with the use of commercial kits (R§D Systems).

The ratio of SFlt1:PIGF will be calculated. All the participants will be followed up at 3 months and 1 year in which blood pressure, UACR and serum creatinine will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* more than 24 weeks of gestation who were diagnosed and classified as preeclampsia or gestational hypertension by the criteria recommends by the American College of Obstetricians and Gynecologists (ACOG)

Severe preeclampsia will be diagnosed by:

* A systolic/diastolic blood pressure ≥ 140 mmHg occurring on two occasions at least 4 hours apart after 20 weeks of gestation a women whose blood pressure has previously been normal
* Proteinuria with excretion of 0.3 gm or more of protein in a 24 hour urine specimen or urine dipstick results of at least 1+(30 mg per deciliter) on two occasions

Exclusion Criteria:

chronic hypertension before pregnancy ,chronic kidney disease according to KDIGO criteria ,twin pregnancies,underlying diabetes mellitus

-

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: pregnant women aged more than 18 years more than 24 weeks of gestation who were diagnosed and classified as preeclampsia or gestational hypertension
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Correlation between serum sFlt-1/PIGF with long term renal function in preeclampsia | 1 year
  measure serum sFlt-1/PIGF and eGFR
Correlation between serum sFlt-1/PIGF with level of blood pressure in preeclampsia | 1 year
  measure serum sFlt-1/PIGF and blood pressure
Correlation between serum sFlt-1/PIGF with level of proteinuria in preeclampsia | 1 year
  measure serum sFlt-1/PIGF and UACR
Correlation between serum endoglin with long term renal function in preeclampsia | 1 year
  measure endoglin and eGFR
Correlation between serum endoglin with blood pressure in preeclampsia | 1 year
  measure endoglin and blood pressure
Correlation between serum endoglin with level of proteinuria in preeclampsia | 1 year
  measure endoglin and UPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Vajira Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] Magee LA, von Dadelszen P. Pre-eclampsia and increased cardiovascular risk. BMJ. 2007 Nov 10;335(7627):945-6. doi: 10.1136/bmj.39337.427500.80. Epub 2007 Nov 1. PMID 17975257
- [Background] Rudra CB, Williams MA. Monthly variation in preeclampsia prevalence: Washington State, 1987-2001. J Matern Fetal Neonatal Med. 2005 Nov;18(5):319-24. doi: 10.1080/14767050500275838. PMID 16390791
- [Background] Vikse BE, Irgens LM, Leivestad T, Skjaerven R, Iversen BM. Preeclampsia and the risk of end-stage renal disease. N Engl J Med. 2008 Aug 21;359(8):800-9. doi: 10.1056/NEJMoa0706790. PMID 18716297
- [Background] McDonald SD, Han Z, Walsh MW, Gerstein HC, Devereaux PJ. Kidney disease after preeclampsia: a systematic review and meta-analysis. Am J Kidney Dis. 2010 Jun;55(6):1026-39. doi: 10.1053/j.ajkd.2009.12.036. Epub 2010 Mar 25. PMID 20346562
- [Background] Khashan AS, Evans M, Kublickas M, McCarthy FP, Kenny LC, Stenvinkel P, Fitzgerald T, Kublickiene K. Preeclampsia and risk of end stage kidney disease: A Swedish nationwide cohort study. PLoS Med. 2019 Jul 30;16(7):e1002875. doi: 10.1371/journal.pmed.1002875. eCollection 2019 Jul. PMID 31361741
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Chaiworapongsa T, Romero R, Kim YM, Kim GJ, Kim MR, Espinoza J, Bujold E, Goncalves L, Gomez R, Edwin S, Mazor M. Plasma soluble vascular endothelial growth factor receptor-1 concentration is elevated prior to the clinical diagnosis of pre-eclampsia. J Matern Fetal Neonatal Med. 2005 Jan;17(1):3-18. doi: 10.1080/14767050400028816. PMID 15804781
- [Background] Venkatesha S, Toporsian M, Lam C, Hanai J, Mammoto T, Kim YM, Bdolah Y, Lim KH, Yuan HT, Libermann TA, Stillman IE, Roberts D, D'Amore PA, Epstein FH, Sellke FW, Romero R, Sukhatme VP, Letarte M, Karumanchi SA. Soluble endoglin contributes to the pathogenesis of preeclampsia. Nat Med. 2006 Jun;12(6):642-9. doi: 10.1038/nm1429. Epub 2006 Jun 4. PMID 16751767
- [Background] Taylor RN, Grimwood J, Taylor RS, McMaster MT, Fisher SJ, North RA. Longitudinal serum concentrations of placental growth factor: evidence for abnormal placental angiogenesis in pathologic pregnancies. Am J Obstet Gynecol. 2003 Jan;188(1):177-82. doi: 10.1067/mob.2003.111. PMID 12548214